CLINICAL TRIAL: NCT05420428
Title: Applying High Resolution Impedance Manometry for Perioperative Swallowing Changes in Older Patients Receiving Endotracheal Intubation or Supraglottic Airway Devices During Orthopedic Surgery: a Pilot Randomized Controlled Trial
Brief Title: Applying High Resolution Impedance Manometry for Perioperative Swallowing Changes in Older Patients Receiving Endotracheal Intubation or Supraglottic Airway Devices During Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202204071RINC
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2022-06

CONDITIONS: Hypopharyngeal Mean Pressure
MeSH Terms: interventions — Laryngeal Masks; Intubation, Intratracheal

STUDY DESIGN:
Intervention Model Description: controll group: tracheal intubation; intervention group: supraglottic airway device
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: We masked the participants, care provider and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endotracheal intubation (Placebo Comparator): under general anesthesia, patients received tracheal intubation.
  Interventions: Device: endotracheal intubation
- supraglottic airway device (Experimental): under general anesthesia, patients received supraglottic airway device
  Interventions: Device: supraglottic airway device

INTERVENTIONS:
Device: supraglottic airway device — under general anesthesia, patients received supraglottic airway device
  Other Names: laryngeal mask airway
  Arms: supraglottic airway device
Device: endotracheal intubation — under general anesthesia, patients received endotracheal intubation
  Arms: endotracheal intubation

SUMMARY:
We aimed to investigate whether patients with tracheal intubation has high hypopharyngeal pressure than patients with supraglottic airway does by using high resolution impedance manometry. We expected that the patients with endotracheal intubation have higher hypopharyngeal pressure than the patients with supraglottic airway devices.

DETAILED DESCRIPTION:
Background: More and more older patients required to receive orthopedic surgery recently. The intubation or supraglottic airway device are required to maintain airway during general anesthesia. Previous studies only reported the subjective swallowing discomfort feeling, however, the objective data was limited. The high-resolution impedance manometry could detect the swallowing muscle power changes with multiple pressure sensors and impedance channels.

Objectives: we aimed to investigate whether patients with tracheal intubation has high hypopharyngeal pressure than patients with supraglottic airway does Patients and methods: The patients receive orthopedic surgery with older than 60 years old. They received high resolution impedance manometry examination at preoperative day, in the post-anesthetic care unit, postoperative day 3 to 7 (pick a day) along with subjective questionnaires. We also followed the IDDSI guideline to test different viscosity of the patients' tolerance for food.

Expected result: The patients with endotracheal intubation have higher hypopharyngeal pressure than the patients with supraglottic airway devices.

ELIGIBILITY:
Inclusion Criteria:

* The patients receive orthopedic surgery with older than 60 years old including 60 years old.

Exclusion Criteria:

* The patients had severe major organ dysfunction

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
hypopharyngeal mean peak pressure | 15 minutes
  hypopharyngeal pressure during food bolus transmittion

CONTACTS AND LOCATIONS:
Locations (1):
- Chih-Min Liu, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
ethical issue